CLINICAL TRIAL: NCT02690597
Title: Validation and Pertinence of Anxiety Analogic Visual Scale in Pain Management by Mobile Acute Pain Team
Brief Title: Validation and Pertinence of Anxiety Analogic Visual Scale in Pain Management
Acronym: ANXYDOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12 560 07; 2013-A00451-44 (Other: France: Agence Nationale de Sécurité du Médicament)
Record Dates: First submitted 2016-02-05; First posted 2016-02-24 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Anxiety; Pain
Keywords: Anxiety analogic visual scale; Pain; State Trait Inventory anxiety scale; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient (Other): State-trait anxiety inventory Y-A form (STAI Y-A form)
  Anxiety visual analog scale evaluation(A-AVS).
  Interventions: Other: Anxiety visual analog scale

INTERVENTIONS:
Other: Anxiety visual analog scale — Anxiety visual analog scale is a test of evaluation of anxiety done by the patient, this scale do not include number and the patient have to place a coloured marker at the level indicating his anxiety feeling

SUMMARY:
Screening of anxiogenic part of pain is an imperative during a medical pain consultation. The actual tools for evaluation of this specific part are complex and time consuming.

To date, it lacked a reliable and reproductive tool to quickly evaluate anxiety of patient in pain. The purpose of this study is to demonstrate the pertinence and validity of anxiety analogic visual scale by comparison with the actual reference the self-assessment questionnaire State Trait Inventory Anxiety Y-A form.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Male or female aged from ≥ 18 years old
* Perfect patient ability to understand and write French
* Patient with a pain threshold permitting a initial medication free consultation and completion of anxiety surveys.

Exclusion Criteria:

* Inability of patient to understand the study procedures and thus inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of pertinence of anxiety analogic visual scale in systematic use as assessed by anxiety levels obtained with State Trait of anxiety Y-A form score | Baseline
  The patient's inclusion take place during the only study participation day of the patient
Evaluation of validity of anxiety analogic visual scale in systematic use as assessed by anxiety levels obtained with State Trait of anxiety Y-A form score | Baseline
  The patient's inclusion take place during the only study participation day of the patient
Evaluation of pertinence of anxiety analogic visual scale in systematic use as assessed by anxiety levels obtained with anxiety analogic visual scale score | Baseline
  The patient's inclusion take place during the only study participation day of the patient
Evaluation of validity of anxiety analogic visual scale in systematic use as assessed by anxiety levels obtained with anxiety analogic visual scale score | Baseline
  The patient's inclusion take place during the only study participation day of the patient

SECONDARY OUTCOMES:
Evaluation of pain consultation impact on anxiety part of pain as assessed by anxiety levels obtained with State Trait of anxiety Y-A form score | Baseline
  The patient's inclusion take place during the only study participation day of the patient
Evaluation of pain consultation impact on anxiety part of pain as assessed by anxiety levels obtained with anxiety analogic visual scale score | Baseline
  The patient's inclusion take place during the only study participation day of the patient
Evaluation of clinical utility of anxiety analogic visual scale in nursing care as assessed by anxiety levels obtained with State Trait of anxiety Y-A form score | Baseline
  The patient's inclusion take place during the only study participation day of the patient
Evaluation of clinical utility of anxiety analogic visual scale in nursing care as assessed by anxiety levels anxiety analogic visual scale score | Baseline
  The patient's inclusion take place during the only study participation day of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe FOISSAC, Nurse, Principal Investigator — CHU Rangueil
Locations (1):
- CHU Rangueil, Toulouse, France

IPD SHARING:
Plan to Share IPD: No